CLINICAL TRIAL: NCT03389022
Title: The Effects of Ketamine on Postoperative Pain After Intraoperative Remifentanil Infusions in Bariatric Surgery
Brief Title: Ketamine for Postoperative Pain in Bariatric Surgery
Acronym: KEPOBA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Greta Kasputytė, MD, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BEC-MF-713
Record Dates: First submitted 2017-12-14; First posted 2018-01-03 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Pain, Postoperative; Bariatric Surgery Candidate
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Treatment1 (Active Comparator): 0,15 mg/kg (LBM) of intravenous pre-incisional single bolus injection of ketamine given for bariatric patients in the operating room.
  Interventions: Drug: Ketamine
- Treatment2 (Active Comparator): 0,3 mg/kg (LBM) of intravenous pre-incisional single bolus injection of ketamine given for bariatric patients in the operating room.
  Interventions: Drug: Ketamine
- Treatment3 (Active Comparator): 0,15 mg/kg (LBM) of intravenous pre-incisional single bolus injection, followed by continuous infusion of 1mg/kg ketamine given for bariatric patients in the operating room.
  Interventions: Drug: Ketamine
- Control (Placebo Comparator): The same amount of intravenous single pre-incisional injection of saline for bariatric patients in the operating room.
  Interventions: Drug: Saline
- Treatment4 (Active Comparator): 0,3 mg/kg (LBM) of intravenous pre-incisional single bolus injection, followed by continuous infusion of 1mg/kg ketamine given for bariatric patients in the operating room.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — 0,15 mg/kg pre-incisional single bolus dose of ketamine in the operating room.
  Other Names: Ketamine hydrochloride
  Arms: Treatment1
Drug: Saline — Intravenous injection given pre-incisional in the operating room.
  Other Names: Sodium chloride
  Arms: Control
Drug: Ketamine — 0,3 mg/kg pre-incisional single bolus dose of ketamine in the operating room.
  Other Names: Ketamine hydrochloride
  Arms: Treatment2
Drug: Ketamine — 0,15 mg/kg pre-incisional single bolus dose of ketamine, followed by continuous infusion of 1 mg/kg in the operating room.
  Other Names: Ketamine hydrochloride
  Arms: Treatment3
Drug: Ketamine — 0,3 mg/kg (LBM) of intravenous pre-incisional single bolus injection, followed by continuous infusion of 1mg/kg ketamine given for bariatric patients in the operating room.
  Other Names: Ketamine hydrochloride
  Arms: Treatment4

SUMMARY:
The aim of this study was to evaluate an effect of pre - incisional single injection of low-dose ketamine on postoperative pain after remifentanil infusion in patients undergoing laparoscopic gastric bypass and gastric plication surgery. Ketamine is an old general anaesthetic. Low doses of it might be used as a adjunct in postoperative analgesia.The investigators expect that the low-dose ketamine reduces postoperative pain after bariatric surgeries.

DETAILED DESCRIPTION:
Effective postoperative pain management enhances early postoperative rehabilitation and may improve outcomes of surgical treatment. New analgetic medications and combinations of these are sought for optimal analgesia with lowest possible incidence of side effects. One of the method of multimodal analgesia is a combination of opioids and adjuvant agents, such as ketamine. To our knowledge, the role of ketamine in the treatment of postoperative pain after bariatric surgeries is poorly researched. The investigators hypothesize that ketamine, acting through the N-methyl-D-aspartate receptor (NMDA) and opioid receptors, provides favourable conditions for adequate post-operative pain management.

ELIGIBILITY:
Inclusion Criteria:

* II or III The American Society of Anesthesiologists (ASA) physical status
* age > 18 years
* bariatric surgery with general remifentanil anesthesia

Exclusion Criteria:

* anamnesis of using opioids for the treatment of chronic pain
* opioid dependence
* younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2015-07-22 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2023-06-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity | On the first postoperative day
  Comparison of pain intensity will be recorded in both groups every 15 min in Post Anesthesia Care Unit (PACU) for 2.5 hours. Postoperative pain was treated with boluses of i.v. morphine (3 mg) at 3 min. intervals on request, if pain intensity exceeded the score of 5 according to the Numeric Pain Rating Scale (NPRS) (0-10). After the transfer of patient's to a regular unit, pain intensity was recorded every 6 hours.
Postoperative morphine requirements | On the first postoperative day
  Postoperative morphine requirements will be recorded in both groups in the PACU for 2.5 hours.

SECONDARY OUTCOMES:
Incidence of side effects | On the first postoperative day
  Incidence of side effects will be recorded in both groups on the first postoperative day.
Patients' satisfaction with postoperative analgesia | On the second postoperative day
  Patients' satisfaction with postoperative analgesia will be recorded in both groups on the second postoperative day.The subject could express their level of satisfaction in five possible levels, from "very satisfied" to "very dissatisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Aurika Karbonskienė, MDPhDAssProf, Study Chair — Lithuanian University of Health Sciences

IPD SHARING:
Plan to Share IPD: No